CLINICAL TRIAL: NCT01311206
Title: Determining Efficacy of a Tolerable Means of Strengthening for Older Adults With Knee Osteoarthritis: Partial Blood Flow Restriction Low Intensity Resistance Training
Brief Title: Low Intensity Resistance Training With Partial Blood Flow Restriction for Quadriceps Strengthening
Acronym: PBFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Neil A. Segal, MD, MS, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 201101711
Record Dates: First submitted 2011-02-22; First posted 2011-03-09 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Knee Osteoarthritis; Symptomatic Knee Osteoarthritis
Keywords: knee osteoarthritis; isokinetic knee extensor strength; quadriceps volume; symptomatic knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBFR (Experimental): Partial Blood Flow Restriction (PBFR) during Low-Intensity Exercise.
  Interventions: Other: partial blood flow restriction
- PBFR control (Active Comparator): Low-Intensity Exercise without partial blood flow restriction.
  Interventions: Other: Low intensity exercise without partial blood flow restriction

INTERVENTIONS:
Other: partial blood flow restriction — Partial Blood Flow Restriction (PBFR) Low-Intensity Exercise: using the Biodex 3 Dynamometer in isotonic mode at 10% (first 3 weeks), 15% (following 3 weeks) and 20% (final 3 weeks) of their 1RM for each side, while receiving PBFR in each exercising limb. The padded belts (65 mm in width and 650 mm in length) of the Kaatsu Master™ PBFR device (Sato Sports Plaza, Tokyo, Japan) will be applied to the proximal thigh as near to the hip joint as is comfortable. Before training each leg, subjects will be seated in a chair where an initial belt pressure of 37-40 mmHg will be applied. The belt then will be iteratively pressurized for 30 seconds and then relaxed for 10 seconds in increments of 20 mmHg from 100 mmHg to the final pressure of 160 mmHg. During exercise, the cuff pressure will be continuously controlled and monitored by the PBFR apparatus
  Arms: PBFR
Other: Low intensity exercise without partial blood flow restriction — Low-Intensity Exercise: using the Biodex 3 Dynamometer in isotonic mode at 10% (first 3 weeks), 15% (following 3 weeks) and 20% (final 3 weeks) of their 1RM for each side in each exercising limb without partial blood flow restriction.
  Arms: PBFR control

SUMMARY:
The objective of the proposed research is to assess the efficacy of an eight-week, efficient and tolerable, low-intensity resistance-training program with concurrent application of partial blood flow restriction (PBFR) for improving quadriceps strength and volume in women with risk factors for incident symptomatic or progressive knee OA. This specific aim will be achieved through a randomized, controlled trial, comparing low intensity training with and without PBFR. There have been numerous reports of exercise interventions in people with knee osteoarthritis. However, this research is novel in that it will be the first to use a low intensity regimen that will minimize forces on the knee while still having the potential to lead to clinically meaningful strength gains in older adults with risk factors for incident symptomatic or progressive knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 45-60
* BMI less than 37 and greater than or equal to 25 kg/m2, or a history of a knee joint injury or surgery, or knee symptoms (pain, aching, or stiffness) on most of the last 30 days, or knee osteoarthritis

Exclusion Criteria:

* Resistance training at any time in the last 3 months prior to study
* 5° malalignment of a knee
* Bilateral knee replacement
* Lower limb amputation
* Lower limb surgery in the last 6 months that affects walking ability or ability to exercise
* Back, hip or knee problems that affect walking ability or ability to exercise
* Unable to walk without a cane or walker
* Unable to ascend at least 2 stairs (to enter our building)
* Inflammatory joint or muscle disease such as rheumatoid or psoriatic arthritis or polymyalgia rheumatica
* Multiple sclerosis
* Known neuropathy
* Self-report of Diabetes
* Currently being treated for cancer or having untreated cancer
* Terminal illness (cannot be cured or adequately treated and there is a reasonable expectation of death in the near future)
* Peripheral Vascular Disease
* History of myocardial infarction or stroke in the last year
* Deep Venous Thrombosis
* Chest pain during exercise or at rest
* Use of supplemental oxygen
* Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
* Staff concern for subject health (such as history of dizziness/faintness or current restrictions on activity)
* Concurrent study participation (such as the MOST study)
* Planning to be away for more than one week during the study

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in isokinetic knee extensor strength after 9-week intervention | Outcome will be measured at week 0 (baseline) and approximately 10 weeks later (after completion of 9-week intervention)
  This outcome will measure efficacy of 9-week intervention.

SECONDARY OUTCOMES:
Change in quadriceps volume assessed by MRI after completion of 9-week intervention | outcome will be measured at week 0 and at approximately week 10 (after completion of 9-week intervention)
  This outcome will measure efficacy of the 9-week intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States